CLINICAL TRIAL: NCT07211113
Title: Exploring Effects of Long-lasting Bicarbonate-Sulfate-Calcium-Magnesium Water Intake on Metabolic Dysfunction-Associated Steatotic Liver Disease (MASLD)-Related Outcomes Via Impacting Intestinal Permeability (IP), IP-related Systemic Inflammation, and Oxidative Stress.
Brief Title: Effects of Long-lasting Bicarbonate-Sulfate-Calcium-Magnesium Water Intake on Metabolic Dysfunction-Associated Steatotic Liver Disease (MASLD)-Related Outcome
Acronym: FonteESSEMASLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Alessandro Federico, Full Professor, University of Campania Luigi Vanvitelli
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0001933/i/2023
Record Dates: First submitted 2025-09-29; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: MASLD - Metabolic Dysfunction-Associated Steatotic Liver Disease
Keywords: Intestinal permeability; MASLD; Systemic inflammation; Mineral water; Oxidative stress

STUDY DESIGN:
Intervention Model Description: Eligible participants will be randomly assigned in a 1:1 ratio into two study arms: 1) Group A: received 400 ml/day of Fonte Essenziale® mineral water, taken every morning on an empty stomach for 12 consecutive months, in addition to a specialist-prescribed controlled nutritional regimen, followed by a 6-month water wash-out period of exclusive controlled nutritional regimen; 2) Group B: followed the same specialist-prescribed controlled nutritional regimen without water supplementation
Who Masked: Investigator
Masking Description: The randomization list was generated using online randomization software (http://www.graphpad.com/quickcalcs/index.cfm) using permuted block list generation (to further reduce sequence predictability). Furthermore, the methods and tools used to generate the sequence were tracked. Regarding allocation concealment, the following criteria were also met: the block size was not disclosed to the investigators enrolling the patients; the investigators recruiting the patients did not know to which group the nex
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): 400 ml/day of Fonte Essenziale® mineral water, taken every morning on an empty stomach for 12 consecutive months, in addition to a specialist-prescribed controlled nutritional regimen, followed by a 6-month water wash-out period of exclusive controlled nutritional regimen
  Interventions: Dietary Supplement: Fonte Essenziale® mineral water
- Group B (No Intervention): Patients receiving the same (of Group A) specialist-prescribed controlled nutritional regimen without water supplementation

INTERVENTIONS:
Dietary Supplement: Fonte Essenziale® mineral water — 400 ml/day of Fonte Essenziale® mineral water, taken every morning on an empty stomach for 12 consecutive months, in addition to a specialist-prescribed controlled nutritional regimen
  Other Names: Bicarbonate-Sulfate-Calcium-Magnesium Water
  Arms: Group A

SUMMARY:
Background: Fonte Essenziale®, a mineral water rich in bicarbonate, sulphate, calcium, and magnesium, has shown potential in modulating the gut-liver axis and microbiota in hepatic steatosis. However, its long-term effects on intestinal permeability (IP), systemic inflammation (SI), and oxidative stress-key factors in Metabolic dysfunction-Associated Steatotic Liver Disease (MASLD) -remain unexplored.

MASLD patients will be consecutively endoller and randomized into two groups: group A receiving Fonte Essenziale® (400 ml/day, fasting) plus a controlled nutritional regimen for 12 months, followed by a 6-month water washout; group B followed only the controlled nutritional regimen. IP markers, SI (IL-1β, IL-6, TNF-α), oxidative stress (dROMs/BAP), and clinical data (including Controlled Attenuation Parameter - CAP) will be assessed at baseline (T0), 12 months (T12), and post-washout (T18). Baseline increased IP (in-IP) was defined by fecal zonulin >110 ng/ml and serum LBPp >10 µg/ml; improvement (im-IP) required normalization of both. A ≥30% CAP reduction will indicate hepatic steatosis improvement.

DETAILED DESCRIPTION:
This will be a prospective, randomized, controlled clinical trial conducted at the Hepatogastroenterology Division of the University of Campania "Luigi Vanvitelli" (Naples, Italy). The study will be designed and implemented under the framework of the Ferrarelle-Vanvitelli research agreement (n. 390-01583577-30059 - dated 09/02/2023), which previously enabled the investigation of mineral water as a non-pharmacological intervention in chronic liver disease.

Patients meeting the diagnostic criteria for MASLD [17] will be consecutively screened for potential eligibility. All individuals considered potentially eligible will undergo Transient Elastography (TE) with Liver Stiffness Measurement (LSM) to exclude those with LSM-defined advanced fibrosis (AF) (> F3).

Eligible participants will then be randomized in a 1:1 ratio into two study arms: Group A and Group B. Group A will receive 400 ml/day of Fonte Essenziale® mineral water, administered each morning on an empty stomach for 12 consecutive months, in addition to a specialist-prescribed controlled nutritional regimen (see dedicated subsection), followed by a 6-month washout period during which only the nutritional regimen will be maintained. Group B will follow the same 12-month nutritional protocol without water supplementation. The selected water dose and fasting administration will be based on the original protocol and prior studies, given that gastric emptying is accelerated and absorption more consistent under fasting conditions, potentially enhancing mucosal interaction.

Three study time-points will be defined: baseline (T0), after 12 months (T12), and post-washout (T18), the latter applicable only to Group A. At each time-point, anthropometric, clinical, and demographic data-including age, sex, smoking status, MASLD-related comorbidities, and Body Mass Index (BMI)-will be collected, alongside routine biochemical parameters and TE-derived liver disease progression metrics, including both LSM-defined fibrosis staging and Controlled Attenuation Parameter (CAP)-based steatosis grading. At T12, a ≥30% reduction in baseline CAP values will be considered indicative of steatosis improvement.

Additionally, at each time-point, following the collection of 20 ml serum and 200 mg fecal samples, intestinal permeability (IP) will be assessed via a biomarker panel comprising fecal zonulin (ng/ml), serum LPS-binding protein (LBPp) (µg/ml), indicative of systemic endotoxin exposure, and serum occludin and claudin-1 (ng/ml), representing epithelial tight-junction integrity. At T0, concurrent fecal zonulin >110 ng/ml and serum LBPp >10 µg/ml will define increased IP (in-IP) [6,13]. At T12, improvement in IP (im-IP) will be defined by simultaneous reductions in fecal zonulin <110 ng/ml and serum LBPp <10 µg/ml. This dual-marker approach will be adopted to enhance diagnostic reliability, as single biomarkers may inadequately reflect barrier integrity and function.

IP-associated systemic inflammation (SI) will be evaluated at all time-points by measuring circulating LPS (ng/ml) and pro-inflammatory cytokines [interleukin (IL)-1β, IL-6, and Tumor Necrosis Factor alpha (TNF-α), pg/ml]. Finally, systemic oxidative stress will be assessed using the Biological Antioxidant Potential (BAP) and derivatives of Reactive Oxygen Metabolites (dROM) tests, both validated tools in chronic liver disease contexts.

ELIGIBILITY:
The inclusion criteria were: age > 18 years, imaging ultrasound-based evidence of hepatic steatosis, and clinical and biochemical features configuring MD (at least one of: obesity, type 2 diabetes, dyslipidemia, or essential arterial hypertension diagnosis).

All patients who were potentially considered eligible received TE evaluation with the LSM definition. Importantly, patients with AF (TE-assessed LSM confirming >F3) were excluded. This choice was motivated by evidence that in AF, IP is significantly altered, contributing to an enhanced bacterial translocation, both events influenced by the potential presence of portal hypertension Other exclusion criteria were: (a) chronic liver disease (CLD) of other etiology [hepatitis B and/or C virus, alcohol-related liver disorder (ALD) with evidence of alcohol abuse history assessed by using the Alcohol Use Disorders Identification Test questionnaire, hemochromatosis, Wilson's disease, or cholestatic liver disorders]; (b) evidence of cancer, including hepatocellular carcinoma (HCC); (c) acute systemic infections; (d) pregnancy; (e) psychological/psychiatric problems potentially invalidating the informed consent and/or conditions impacting the ability to adhere to dietary recommendations and intervention protocol; (f) chronic kidney disease (with Estimated Glomerular Filtration Rate - eGFR- <30 ml/min); (g) the use (ongoing and/or in the 3 months preceding the enrollment) of drugs/supplements that could influence IP (e.g., probiotics, antibiotics, NSAIDs).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2023-01-29 (Actual); Primary Completion 2025-05-25 (Actual); Study Completion 2025-09-02 (Actual)

PRIMARY OUTCOMES:
Intestinal permeability changes | T0-T12 (after the 12 months of intervention)
  Improving increased intestinal permeability (IP) in group A compared with group B
  Primary End-point (composite):
  Statistically significant reduction of fecal zonulin, simultaneously with a significant increase occludin and claudin 1 serum levels, in group A (compared with group B)
  Note: In each patient, the simultaneous reduction of fecal zonulin (< 110 ng/ml) and serum LPBp (< 10 microg/ml) defined an improvement in IP (i-IP).
Impacting on intestinal permeability | After the 12 months of intervention
  Improving increased intestinal permeability (IP) in group A compared with group B Endpoint: Statistically significant reduction of fecal zonulin, simultaneously with a significant increase occludin and claudin 1 serum levels, in group A (compared with group B)
  Note:In each patient, the simultaneous reduction of fecal zonulin (< 110 ng/ml) and serum LPBp (< 10 microg/ml) defined an improvement in IP (i-IP).

SECONDARY OUTCOMES:
Impacting on altered Intestinal Permeability-related systemic inflammation | T0-T12 (after the 12 months of intervention)
  Improving systemic chronic inflammation status in group A compared with group B , as well as in patients of group A presenting improved IP, compared with those not reaching this outcome
  Secondary End-point:
  Statistically significant reduction of IL-1, TNF-a, IL-6, LPS serum levels in group A (compared with group B), as well as in patients of group A presenting improved IP, compared with those not reaching this outcome
Impacting on clinical outcomes | T0-T12 (after 12 months-intervention)
  Improving hepatic steatosis severity and metabolic features in group A compared with group B, as well as in patients of group A presenting improved IP, compared with those not reaching this outcome
  End-point: Statistically significant reduction of CAP levels in group A (compared with group B), as well as in patients of group A presenting improved IP, compared with those not reaching this outcome
  End-point: Statistically significant reduction of FPG, insulin, TG levels, and increase in HDL serum levels in group A (compared with group B), as well as in patients of group A presenting improved IP, compared with those not reaching this outcome

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Federico, Principal Investigator — University of Campania Luigi Vanvitelli
Locations (1):
- University of Campania Luigi Vanvitelli, Napoli, Campania, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dallio M, Romeo M, Di Nardo F, Senese G, Silvestrin A, Coppola A, Napolitano C, Vaia P, Basile C, Martinelli G, Gregorio A, Federico A. Beneficial Effects of Long-Lasting Bicarbonate-Sulfate-Calcium-Magnesium Water Intake on Metabolic Dysfunction-Associated Steatotic Liver Disease (MASLD)-Related Outcomes via Impacting Intestinal Permeability (IP), IP-Related Systemic Inflammation, and Oxidative Stress. Nutrients. 2025 Oct 31;17(21):3452. doi: 10.3390/nu17213452. PMID 41228524